CLINICAL TRIAL: NCT06790381
Title: Effect of Biological Sex on Multimodal Biomarkers of Disease Progression in Patients with Parkinson's Disease: from Pathophysiological Mechanisms to Equitable Health Outcomes
Brief Title: Effect of Biological Sex on Multimodal Biomarkers of Disease Progression in Patients with Parkinson's Disease
Acronym: GENDERIZE-PD
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Università della Campania Luigi Vanvitelli (Unknown); University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, FULL PROFESSOR, IRCCS San Raffaele
Other Study IDs: GENDERIZE-PD
Record Dates: First submitted 2025-01-10; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: sex Hormones; Neuroimaging; Biomarkers; Parkinson's Sex differences; Parkinson's progression; non-motor symptoms; motor symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Patients with Parkinson's Disease
- controls: Healthy controls

SUMMARY:
The GENDERIZE-PD study is a research project to understand how biological sex affects the progression of Parkinson's disease (PD). PD is a brain disorder that causes both movement and non-movement symptoms. Researchers aim to identify differences between men and women in how the disease progresses and in the biomarkers (biological indicators) related to the condition.

Study Goals:

Identify differences by sex in how PD develops and progresses, using clinical assessments, brain scans, and blood tests.

Find predictors of disease progression that may help create personalized treatments for men and women.

Study Details:

Type of Study: Observational, with additional procedures (e.g., blood tests and brain scans).

Participants:

120 people with early-stage PD (60 men, 60 women) diagnosed within the last 3 years.

90 healthy participants (caregivers or relatives) for comparison.

Procedures:

Clinical exams and questionnaires about movement and non-movement symptoms (like sleep, mood, and fatigue).

Blood tests to measure hormone levels. Brain imaging to study changes in structure and activity. Timeline: Participants will be followed for 18 months, with evaluations at 0, 6, 12, and 18 months.

Why This Study is Important:

Men and women often experience PD differently. For example:

Men are more likely to have memory and thinking problems. Women may develop movement side effects from treatments more often.

Understanding these differences can lead to:

Improved care plans tailored to men and women. Better treatment outcomes by focusing on sex-specific factors.

Who Can Join:

Adults aged 18-80 with early-stage PD or healthy individuals willing to provide blood samples and undergo brain imaging.

Exclusions include women not in menopause and people with certain medical or other health conditions.

Study Locations:

The study is conducted at three centers in Italy:

San Raffaele Scientific Institute - Milan (led by Prof. Federica Agosta). University of Campania "Luigi Vanvitelli" - Naples (led by Prof. Alessandro Tessitore).

University "Magna Graecia" - Catanzaro (led by Prof. Gennarina Arabia).

DETAILED DESCRIPTION:
Overview:

The GENDERIZE-PD study investigates how biological sex influences the progression of Parkinson's disease (PD). This groundbreaking project seeks to uncover sex-specific differences in clinical symptoms, disease progression, and biomarkers to enable more personalized and equitable treatment strategies for men and women. By examining a range of biological, clinical, and imaging data, the study aims to provide a deeper understanding of the disease and identify predictors of progression.

Background and Rationale:

PD is a progressive neurodegenerative disorder characterized by motor symptoms (e.g., tremors, rigidity) and non-motor symptoms (e.g., mood disturbances, sleep problems). The disease affects men nearly twice as often as women, and differences between the sexes have been observed in clinical presentations and treatment responses:

* Men with PD are more likely to experience cognitive decline.
* Women with PD are at higher risk of treatment-related motor complications.

Emerging evidence suggests that biological sex impacts brain structure and function, potentially influencing the course of neurodegenerative diseases like PD. Hormonal factors, such as testosterone and estrogen, play key roles in brain health and disease susceptibility. This study seeks to clarify these sex-based differences by analyzing clinical, biological, and neuroimaging data.

Objectives:

The study is designed to achieve the following:

1. Primary Objective: Identify clinical differences between men and women with early-stage PD, focusing on motor and non-motor symptoms, and correlate these findings with sex hormone levels.
2. Secondary Objectives: Investigate sex-specific differences in brain imaging results, including MRI and dopamine transporter (DAT) scans, and biomarker profiles.
3. Exploratory Objectives: Evaluate the predictive value of biomarkers for disease progression and explore sex-independent patterns of PD progression.

Study Design:

This is a multicenter, observational, prospective, case-control study with a longitudinal follow-up of 18 months. The research involves three Italian centers:

1. San Raffaele Scientific Institute - Milan
2. University of Campania "Luigi Vanvitelli" - Naples
3. University "Magna Graecia" - Catanzaro

Study Phases:

1. Baseline Cross-Sectional Analysis: Collect clinical, imaging, and biological data to establish sex-specific profiles at the onset of the study.
2. Longitudinal Follow-Up: Monitor participants over 18 months to track disease progression and evaluate changes in biomarkers.

Participants:

* Total Enrollment: 210 participants.
* 120 individuals with early-stage PD (60 men, 60 women).
* 90 healthy controls (45 men, 45 women).
* Inclusion Criteria: Participants aged 18-80 years with idiopathic early-stage PD (diagnosed within 3 years), Hoehn & Yahr stage ≤2.5, or healthy individuals without neurological disorders.
* Exclusion Criteria: Conditions such as major depression, dementia, or premenopausal status (for women).

Procedures:

Participants will undergo:

* Clinical Assessments: Evaluations of motor (e.g., MDS-UPDRS) and non-motor symptoms (e.g., sleep, mood, fatigue scales).
* Blood Tests: Analysis of hormone levels (e.g., testosterone, SHBG) and calculation of the Free Androgen Index.
* Neuroimaging:
* MRI: Examine structural and functional changes in the brain.
* DAT Scans: Assess dopamine transporter binding levels.
* Questionnaires and Interviews: Assess emotional well-being, cognitive function, and quality of life.

Outcome Measures:

* Primary Outcomes: Sex-related differences in clinical and biomarker profiles at baseline and follow-up.
* Secondary Outcomes: Correlations between neuroimaging findings and clinical measures.
* Exploratory Outcomes: Biomarker trajectories over time and their predictive value for disease progression.

Significance:

This study addresses critical gaps in understanding sex-based differences in PD. By integrating clinical, biological, and imaging data, the results could:

* Improve understanding of PD's natural history.
* Highlight the importance of considering sex as a factor in research and treatment design.
* Lead to more personalized and equitable healthcare strategies.

Funding and Ethical Considerations:

The study is funded by the European Union's NextGenerationEU initiative and the Italian Ministry of University and Research (PRIN). It adheres to the Declaration of Helsinki, Good Clinical Practice guidelines, and all relevant regulatory standards. Written informed consent will be obtained from all participants before enrollment.

Implications for Future Research:

Findings from the GENDERIZE-PD study will inform the design of sex-specific clinical trials and potentially contribute to the development of disease-modifying therapies. By considering sex as a key biological variable, this research aims to set a new standard for inclusivity and precision in PD care.

ELIGIBILITY:
Inclusion Criteria:

Patients with Parkinson's Disease:

* Age: 18-80 years old
* Idiopathic early-stage Parkinson's Disease (≤3 years of disease)
* Stage ≤2.5 on the Hoehn&Yahr scale Able to give informed consent

Healthy controls:

-Age: 18-80 years old Able to give informed consent

Exclusion Criteria:

* Patients with Parkinson's Disease:
* Presence of Parkinson's Disease dementia
* Presence of major depression or other dysthymic disorders according to DSM-IV criteria
* Women not in menopause (menopause is a point in time 12 months after a woman's last period)
* Any other relevant neurological or medical condition

Healthy controls:

* Women not in menopause (menopause is a point in time 12 months after a woman's last period)
* Any other relevant neurological or medical condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease and healthy controls
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
MDS-sponsored revision of the Unified Parkinson's Disease Rating Scale | 0,6,12, 18 months
  The International Parkinson and Movement Disorder Society sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a comprehensive 50 question assessment of both motor and non-motor symptoms associated with Parkinson's

SECONDARY OUTCOMES:
Sex hormones (free androgens index) | Baseline, 12 months
  In this study we will measure levels of testosterone and sex hormones binding protein (SHBG). Blood samples (5ml) from all subjects will be taken between 8 and 10 a.m. in the supine position after a 30-min rest. The hormone concentrations will be measured using chemiluminescent reactions. Using these results, free androgens index (FAI) will be evaluated (by dividing total testosterone level by the SHBG level and multiplying by 100). B2 will be collected in both patients with PD and controls at T0 and T12 visits.

OTHER OUTCOMES:
Magnetic resonance imaging | 0,12 months
  Structural MRI. 3D T2-weighted and fluid-attenuated inversion recovery (FLAIR) images will be acquired to exclude CNS lesions, while T1-weighted sequences will assess grey matter alterations. T1-weighted imaging will be used to analyze cortical thickness and grey matter volume in cortical and subcortical regions of PD patients. Structural MRI analysis includes cortical thickness evaluation, voxel-based morphometry, and regional grey matter volume assessment.
  Diffusion Tensor Imaging (DTI) metrics will assess microstructural white matter damage in PD. Resting-state fMRI (RS-fMRI). RS-fMRI evaluates brain networks and their functional interplay. Connectivity will be analyzed for motor/non-motor networks and striatal subregions. Gender-specific differences will also be explored. Graph-based network analysis represents the state-of-the-art methodology to assess brain connectivity.
(123)I-2β-carbomethoxy-3β-(4-iodophenyl)-N-(3-fluoropropyl)-nortropane ((123)I-FP-CIT) SPECT. | baseline
  123I-FP-CIT SPECT acquisition and processing procedures will be performed according to the European Association. Patients will receive perchlorate (1,000 mg) 30 min before scanning to block thyroid uptake of free radioactive iodine. Brain imaging will be performed 3 hours after the administration of 200 MBq of 123I-ioflupane (GE-Amersham, Eindhoven, The Netherlands) using a dual-headed gamma camera (Infinia Hawkeye; General Electric, Milwaukee, WI) equipped with low-energy, high-resolution collimators. Scans will be acquired with a photopeak window centered on 159 keV 610% with a 128 3128 image matrix (zoom factor: 1.5; 40 s per view and 2 3 64 views). Patients will be carefully positioned in the gamma camera, with their meato-orbital axis in a transverse plane to reduce reorientation during reconstruction, in a special head holder that allows a minimal rotation distance. Images will be reconstructed using filtered back projection with a Butterworth filter (cut-off 0.5 and order 6). T
Unified Dyskinesia Rating Scale (UDysRS) | 0,6,12,18 months
  The Unified Dyskinesia Rating Scale captures the essential features of dyskinesia in Parkinson's disease within a single scale, including patient perceptions, time factors, anatomical distribution, objective impairment, severity, and disability. The scale addresses the issues clinically pertinent to physicians dealing with dyskinesia in clinical and research settings as well as the issues clinically pertinent to patients experiencing dyskinesia
Freezing of Gait Questionnaire (FOGq) | 0,6,12,18 months
  The FOGQ assesses Freezing of Gait (FOG) severity unrelated to falls in patients with Parkinson's Disease (PD), FOG frequency, disturbances in gait, and relationship to clinical features conceptually associated with gait and motor aspects (e.g., turning).
Nonmotor Symptom assessment scale for PD (NMSS) | 0,6,12,18 months
  The Non-Motor Symptoms Scale (NMSS) is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions. The scale can be used for patients at all stages of PD.
Apathy evaluation scale (AES) | 0, 12 months
  The Apathy Evaluation Scale (AES) is a tool utilized with individuals with brain injury, neurocognitive disorders, and other mixed populations, to quantify and characterize apathy in adults.The scale "treats apathy as a psychological dimension defined by simultaneous deficits in the overt behavioral, cognitive, and emotional concomitants of goal-directed behavior."
Parkinson Anxiety Scale (PAS) | 0,12 months
  The Parkinson's disease (PD)-specific Parkinson Anxiety Scale (PAS) is an anxiety rating scale that has been validated in cross-sectional studies.
Beck Depression Inventory (BDI) | 0,12 months
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.
Parkinson's Disease Sleep Scale (PDSS) | 0,12 months
  The PDSS is a reliable, valid, precise, and potentially treatment-responsive tool for measuring sleep disorders in PD
Parkinson's Disease Fatigue Scale (PFS) | 0,12 months
  The PFS is a patient rated scale that reflects the physical aspects of fatigue in patients with Parkinson's Disease
Barratt Impulsiveness Scale-11 (BIS-11) | 0, 12 months
  The Barratt Impulsiveness Scale (BIS-11) is a widely utilized 30-item self-report instrument for assessing impulsivity.
Temperament and Character Inventory (TCI) | 0, 12 months
  The Temperament and Character Inventory (TCI) is a widely used self-report measure of personality.
Questionnaire for impulsive-compulsive disorders in Parkinson's disease Rating Scale (QUIP-RS) | 0,12 months
  the QUIP-RS is valid and reliable as a rating scale for ICDs and related behaviors reported to occur in PD patients
Assessment of Autonomic Dysfunction in Parkinson's Disease (SCOPA-AUT) | 0, 12 months
  The SCOPA-AUT was developed to evaluate autonomic symptoms in patients with Parkinson's disease. The scale is self-completed by patients and consists of 25 items assessing the following domains: gastrointestinal (7), urinary (6), cardiovascular (3), thermoregulatory (4), pupillomotor (1), and sexual (2 items for men and 2 items for women).
King's PD Pain Scale (KPPS) | 0,12 months
  The KPPS is an evaluative measure for pain-related symptoms in PD with "lumping" of various types of pain symptoms together.
REM Sleep Behavior Disorder Single Question (RBDSQ) | 0, 12 months
  The REM Sleep Behavior Disorder Single-Question Screen (RBD1Q) is a one-question screening tool for dream enactment behaviors associated with the parasomnia REM sleep behavior disorder (RBD). It screens for RBD with a simple yes/no response.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Agosta, MD,PhD, Principal Investigator — IRCCS San Raffale, Milan

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data that underlie published results may be shared with qualified researchers upon request, in accordance with applicable ethical and legal guidelines.